CLINICAL TRIAL: NCT00147251
Title: Stop Atherosclerosis in Native Diabetics Study
Acronym: SANDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cynthia West (Other)
Responsible Party: Sponsor-Investigator, Cynthia West, Phoenix Field Office Manager, Medstar Health Research Institute
Organization: Medstar Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000-285; Grant # 1 U01 HL67031 (Other Grant/Funding Number: NHLBI); NCT00047424 (obsolete NCT alias)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Disease; Hypertension; Hyperlipidemia; Diabetes; Carotid Atherosclerosis
Keywords: lowering LDL and BP below current targets; LDL cholesterol treatment; blood pressure treatment; carotid intimal medial thickness; prevent progression of CVD
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias; Diabetes Mellitus; Carotid Artery Diseases | interventions — Cholesterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SANDS Control Group (No Intervention): Standard Treatment for blood pressure and cholesterol
- SANDS Intervention Group (Active Comparator): FDA approved drugs to treat blood pressure and cholesterol
  Interventions: Drug: FDA approved drugs to treat blood pressure and cholesterol

INTERVENTIONS:
Drug: FDA approved drugs to treat blood pressure and cholesterol
  Other Names: No Intervention
  Arms: SANDS Intervention Group

SUMMARY:
Compared to standard treatment goals achieving lower targets for LDL cholesterol (bad cholesterol) and blood pressure in people with diabetes will slow the progression of atherosclerosis as measured by carotid artery thickness, and reduce clinical cardiovascular events such as heart attacks and strokes. This study is a randomized 3-year trial. The primary endpoint will be a combination of various measures of the carotid artery, (which is an easy, non-invasive way to detect cardiovascular disease) and events such as heart attacks and strokes. The study will also look at secondary endpoints such as how well the heart pumps, fat,protein and inflammatory markers in the blood,and kidney function. The study enrolled 549 American Indian men and women with diabetes, > 40 years of age and is being conducted in four field centers involving Indian Health Service/Tribal primary care facilities in Phoenix/Sacaton, Arizona; Chinle, Arizona; Rapid City/Pine Ridge, South Dakota; and Lawton, Oklahoma, with input from American Indian physicians and community members.

DETAILED DESCRIPTION:
Diabetes incidence is increasing rapidly in the United States. Diabetes increases the risk for CVD, the major cause of death in diabetic individuals. The conventional cardiovascular risk factors of hyperlipidemia and hypertension add to the progression of diabetic vascular disease. Appropriate treatment targets for LDL-C and blood pressure in diabetic individuals are currently being debated. The Stop Atherosclerosis in Native Diabetics Study is a randomized, open label, 3-year, clinical trial to examine the effects of aggressive LDL-C (goal < 70 mg/dL) and BP (goal < 115/75 mm Hg) reduction versus the standard goals of < 100 mg/dL for LDL-C and < 130/85 mmHg for BP. Five hundred forty-nine American Indian men and women > age 40 with type 2 diabetes were randomized to one of two groups. Lipids and BP are managed using FDA-approved medications in an algorithmic approach. The presence and progression of atherosclerosis are evaluated by carotid ultrasonography; echocardiography assesses cardiac function. The primary endpoint is the composite outcome of change in carotid artery intimal medial thickness and fatal/nonfatal cardiovascular events. These outcomes are combined by using a ranked analysis for carotid thickness and assigning a "worst rank" for a cardiovascular event. Secondary endpoints include carotid plaque score, left ventricular geometry and function, serum CRP, and safety measures. Unique aspects of the study design and analysis plan involve changes during the trial of LDL-C treatment goals for participants with baseline or incident CVD in the conventional group, because of changes in the standard of care, and the use of a composite outcome. Study results will be valuable in understanding the effects of aggressive risk factor reduction on atherosclerosis burden and cardiac function in diabetic individuals in all U.S. populations and will provide evidence for determining optimal LDL-C and BP treatment goals for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. American Indian men and women 40 years of age or older
2. Type 2 DM (according to 1997 ADA criteria and/or previously diagnosed by former ADA or WHO criteria): fasting plasma glucose >= 7.0 mmol/L (126 mg/dL) or 2-hour glucose >= 11.0 mmol/L (>200 mg/dL) after a 75-gram oral glucose tolerance test.
3. LDL cholesterol >= 100 mg/dL. within the previous 12 months.
4. Systolic BP >= 130 mm Hg. within the previous 12 months.

Exclusion Criteria:

1. New York Heart Association Stage III- IV congestive heart failure.
2. SBP >180 mmHg (2% of population) or patients with known causes of hypertension.
3. History of angioedema.
4. Any medical condition that study physicians believe would interfere with study participation or evaluation of results.
5. Mental incapacity and/or cognitive impairment on the part of the patient that would preclude adequate understanding of, or cooperation with, the study protocol.
6. Serum hepatic transaminase levels 2X the upper limit of normal.
7. Participation in any clinical trial of any investigational medication within 3 months prior to this trial.
8. Renal insufficiency as indicated by serum creatinine >2.0 for women and >2.4 for men.
9. Diagnosis of primary hyperlipidemia in medical record.
10. Secondary hypercholesterolemia due to hypothyroidism or nephrotic syndrome. Patients on stable doses of thyroid replacement therapy will be eligible.
11. Presence of malignancy or history of any cancer except skin cancer within the past 5 years.
12. Pregnancy or lactation. Premenopausal women will be requested to use birth control methods throughout the study and provided educational materials about the risks of using the study medications during pregnancy.
13. Unable to obtain quantifiable carotid measure during screening examination.
14. Concomitant long term use of cyclosporins (Sandimmune), macrolide antibiotics (erythromycin -many generic and brand name forms, clarithromycin, Biaxin, and Zithromax), azole antifungals (itraconazole-Sporanox, ritonavir, Norvir, and nelfinavir (Viracept).
15. Orthostatic hypotension as defined by the following:

    1. The individual has a measured fall of >20 mmHg in systolic BP upon standing associated with symptoms lasting more than one minute (or severe symptoms that would not allow further lowering of BP)
    2. The standing systolic blood pressure is less than 90 mm.
16. Triglyceride level >350 mg/dl.
17. Severe aortic stenosis with valve area <=1.0 square cm.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2003-05; Primary Completion 2006-11 (Actual); Study Completion 2007-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara V Howard, PhD, Principal Investigator — Medstar Health Research Institute
Locations (4):
- United States (4):
  - Chinle Comprehensive Health Care, Chinle, Arizona
  - Phoenix Indian Medical Center, Phoenix, Arizona
  - USPHS Indian Hospital, Lawton, Oklahoma
  - Black Hills Center for American Indian Health, Rapid City, South Dakota

REFERENCES:
- [Derived] Roman MJ, Howard BV, Howard WJ, Mete M, Fleg JL, Lee ET, Devereux RB. Differential impacts of blood pressure and lipid lowering on regression of ventricular and arterial mass: the Stop Atherosclerosis in Native Diabetics Trial. Hypertension. 2011 Sep;58(3):367-71. doi: 10.1161/HYPERTENSIONAHA.111.172486. Epub 2011 Jul 25. PMID 21788602
- [Derived] Fleg JL, Mete M, Howard BV, Umans JG, Roman MJ, Ratner RE, Silverman A, Galloway JM, Henderson JA, Weir MR, Wilson C, Stylianou M, Howard WJ. Effect of statins alone versus statins plus ezetimibe on carotid atherosclerosis in type 2 diabetes: the SANDS (Stop Atherosclerosis in Native Diabetics Study) trial. J Am Coll Cardiol. 2008 Dec 16;52(25):2198-205. doi: 10.1016/j.jacc.2008.10.031. PMID 19095139
- [Derived] Howard BV, Roman MJ, Devereux RB, Fleg JL, Galloway JM, Henderson JA, Howard WJ, Lee ET, Mete M, Poolaw B, Ratner RE, Russell M, Silverman A, Stylianou M, Umans JG, Wang W, Weir MR, Weissman NJ, Wilson C, Yeh F, Zhu J. Effect of lower targets for blood pressure and LDL cholesterol on atherosclerosis in diabetes: the SANDS randomized trial. JAMA. 2008 Apr 9;299(14):1678-89. doi: 10.1001/jama.299.14.1678. PMID 18398080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified from the local Indian hospital service center, or DM clinic. In March 2004, the DSMB recommended and the SC voted to over-recruit by 10-20% to compensate for the possible need for more aggressive treatment for participants with baseline CVD. Randomization concluded in July 2004 with 547 randomized participants.
Pre-assignment Details: Sonogram eligibility was confirmed by tape review at the core lab prior to randomization. A potential participant had to have LDL-C > 100 mg/dL and systolic BP > 130/85 mmHg. A participant could undergo a maximum of four screening visits within a 3-month period to confirm eligibility.
Groups:
- Standard Treatment: standard targets of LDL-C < 100 mg/dL and BP < 130/85 mm Hg
- Aggressive Treatment: /aggressive targets of LDL-C < 70 mg/dL plus BP < 115/75 mm Hg
Period: Recruitment and Enrollment
Arm/Group | Standard Treatment | Aggressive Treatment
Started | 271 | 277
Completed | 247 | 252
Not Completed | 24 | 25
Not completed — change in treatment guidelines | 24 | 25
Period: Follow up
Arm/Group | Standard Treatment | Aggressive Treatment
Started | 247 | 252
Completed | 247 | 252
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Aggressive Treatment | Total
Number analyzed (Participants) | 247 | 252 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (4.24) | 55.3 (4.24) | 56.1 (4.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 164 | 327
  Male | 84 | 88 | 172

OUTCOME MEASURES:

1. Primary Outcome: Changing LDL Cholesterol
Description: LDL cholesterol intervention to lower targets than are currently recommended to retard atherosclerosis measured by LDL-C mg/dL.
  Scale: LDL cholesterol levels should be less than 100 mg/dL
Time Frame: 36 months
Population: Native American
Measure: Median (Standard Deviation); unit: Mg/dl
Groups:
- Standard Treatment: standard targets of LDL-C < 100 mg/dL and
- Aggressive Treatment: /aggressive targets of LDL-C < 70 mg/dL
Arm/Group | Standard Treatment | Aggressive Treatment
Number analyzed (Participants) | 247 | 252
Mg/dl | 100 (74) | 70 (91)

2. Secondary Outcome: Changing Blood Pressure
Description: Treatment of blood pressure to prevent/reduce diseases of heart and blood vessels. Measured by mmHG.
  Normal values should be below 120/80 mm Hg.
Time Frame: 36 month follow-up
Population: American Indian
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- SANDS Control Group: Standard Treatment for blood pressure
- SANDS Intervention Group: FDA approved drugs to treat blood pressure
Arm/Group | SANDS Control Group | SANDS Intervention Group
Number analyzed (Participants) | 247 | 252
mm Hg | 130 (.001) | 115 (.001)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | SANDS Control Group | SANDS Intervention Group
Serious Adverse Events (participants affected / at risk) | 1/247 | 4/252
Other Adverse Events (participants affected / at risk) | 0/247 | 0/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SANDS Control Group (N=247) | SANDS Intervention Group (N=252)
Heart Attack (Vascular disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No